CLINICAL TRIAL: NCT00160264
Title: A Randomized, Double-Blind, Multicenter, Parallel Pilot Clinical Trial to Study the Efficay of a Treatment of Lactulose + Vitamin D + Calcium 0.5 g Concurrently Controlled With a Standard Treatment (Vit D + Calcium) in Bone Mass Preservation Among Postmenopausal Women
Brief Title: Study to Investigate if Adding Lactulose to Vitamin D and Calcium Has an Effect on the Preservation of Bone in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: S105.4.107
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Osteopenia
Keywords: lactulose; randomised clinical trial; osteopenia; postmenopause
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Lactulose; Vitamin D; Calcium

INTERVENTIONS:
Drug: Lactulose, Vitamin D, Calcium

SUMMARY:
This is a randomized, double-blind, multicentre, parallel pilot clinical trial to study the efficacy of a treatment of lactulose 15 ml + vitamin D 400 U + calcium 0.5 g compared to lactulose placebo 15 ml + vitamin D 400 U + calcium 1 g in bone mass preservation among postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 55 and 65 years old; postmenopausal who have amenorrhea for 5 or more years; women with the diagnosis of osteopenia defined DMO -1,5 to -2,5

Exclusion Criteria:

Any disease causing osteopenia (hyperthyroidism, hyperparathyroidism, hypercortisolism, osteogenesis imperfecta, rheumatoid arthritis, homocystinuria, etc.)

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-01

PRIMARY OUTCOMES:
bone mass preservation by bone densitometry values in 1 year period

SECONDARY OUTCOMES:
evolution of bone remodelling parameters

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (3):
- Spain (3):
  - Site 1, Barcelona
  - Site 2, Barcelona
  - Site 3, Barcelona